CLINICAL TRIAL: NCT04262804
Title: A Randomized, Open-Label, Multiple-center, Phase II Study to Evaluate the Efficacy and Safety of Margetuximab Plus Chemotherapy vs Trastuzumab Plus Chemotherapy in the Treatment of Chinese Patients With HER2+ Metastatic Breast Cancer Who Have Received Prior Anti-HER2 Therapies
Brief Title: A Study to Evaluate the Efficacy and Safety of Margetuximab Plus Chemotherapy in the Treatment of Chinese Patients With HER2+ MBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1302-002
Record Dates: First submitted 2020-01-30; First posted 2020-02-10 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer Metastatic
Keywords: Breast Cancer Metastatic; MBC; Margetuximab
MeSH Terms: interventions — margetuximab; Trastuzumab; Capecitabine; Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Margetuximab & Chosen Chemotherapy (Experimental): The dosage and administering of margetuximab is 15 mg/kg IV every 21 days. Investigators need to chose one of the 3 chemotherpies based on patient conditions.
  Interventions: Drug: Margetuximab; Drug: Chosen Chemotherapy (Capecitabine); Drug: Chosen Chemotherapy (Vinorelbine ); Drug: Chosen Chemotherapy (Gemcitabine )
- Trastuzumab & Chosen Chemotherapy (Active Comparator): The dosage and administering of Trastuzumab is 8 mg/kg loading dose then 6 mg/kg IV every 21 days. Investigators need to chose one of the 3 chemotherpies based on patient conditions.
  Interventions: Drug: Trastuzumab; Drug: Chosen Chemotherapy (Capecitabine); Drug: Chosen Chemotherapy (Vinorelbine ); Drug: Chosen Chemotherapy (Gemcitabine )

INTERVENTIONS:
Drug: Margetuximab — Margetuximab IV
  Arms: Margetuximab & Chosen Chemotherapy
Drug: Trastuzumab — Trastuzumab IV
  Arms: Trastuzumab & Chosen Chemotherapy
Drug: Chosen Chemotherapy (Capecitabine) — Capecitabine tablet
Drug: Chosen Chemotherapy (Vinorelbine ) — Vinorelbine IV
Drug: Chosen Chemotherapy (Gemcitabine ) — Gemcitabine IV

SUMMARY:
This is a randomized, open-label, multi-center, Phase II clinical study to evaluate the efficacy and safety of margetuximab plus chemotherapy compared with trastuzumab plus chemotherapy in Chinese patients (Mainland, Hong Kong and Taiwan) with advanced HER2+ breast cancer who have received at least 2 prior lines of anti-HER2 directed therapy in the metastatic setting (mandatory including trastuzumab).

The primary endpoint of this study is PFS evaluated by BICR. The secondary endpoints are OS, PFS evaluated by investigator, ORR, DoR, CBR, safety and tolerability, the impact of ADA, and the popPK profile

DETAILED DESCRIPTION:
Approximately 120 Chinese subjects will be enrolled and randomized to treatment group and control group in 1:1 fashion, approximately 60 subjects in each group. Eligible subjects are HER2 positive, metastatic breast cancer who has received at least 2 prior lines of anti-HER2 directed therapy in the metastatic setting (mandatory to have trastuzumab, and other anti-HER2 agents e.g. lapatinib, pyrotinib, and pertuzumab; in case of having received (neo)adjuvant anti-HER2 therapy) in Chinese patients (Mainland, Hong Kong and Taiwan). Subjects should Have received treatment with at least one, and no more than three, lines of therapy overall in the metastatic setting (including anti-HER2 directed therapy and chemotherapy, and patients must have progressed on or following, the most recent line of therapy, based on RECIST 1.1.

Eligible subjects will be randomized 1:1 to receive margetuximab plus chemotherapy compared with trastuzumab plus chemotherapy. The dosage and administering of margetuximab is 15 mg/kg IV Q3W. Trastuzumab was administered 8 mg/kg loading dose, 6 mg/kg subsequent doses, IV Q3W. Prior to randomization to either margetuximab or trastuzumab, investigators selected one of four backbone chemotherapy regimens given at standard doses: capecitabine, vinorelbine or gemcitabine. Capecitabine and vinorelbine should be selected in priority. Gemcitabine could be selected only if capecitabine and vinorelbine were used in previous treatment. Subject will receive the treatment until disease progression, unacceptable toxicity, withdrawal of consent, initiation of subsequent anti-tumor treatment therapy, or death (whichever occurs first). Subject is not allowed to crossover after disease progression. Randomization was stratified by number of metastatic sites (≤2, >2) and chemotherapy chosen.

The definition of HER2 positive is to have at least once 3+ by IHC, FISH positive or CISH positive in the pathological test/retesting. Subject should provide original biopsy/surgical excision tissue sample/latest follow-up sample after randomization, for the centralized test and review when necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to performing any protocol-related procedures
2. Male or female, age ≥ 18 years old at the time of screening.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Subject has histologically confirmed HER2 positive metastatic breast cancer. Note: the definition of HER2 positive is to have at least once 3+ by IHC, FISH positive and CISH positive in the pathological test/retesting conducted at least once by investigational site or qualified central lab which met national standard.
5. Have received at least 2 prior lines of anti-HER2 directed therapy in the metastatic setting (mandatory to have trastuzumab, and other anti-HER2 agents e.g. lapatinib, pyrotinib, pertuzumab, or T-DM1), regardless of having received (neo)adjuvant anti-HER2 therapy or not
6. Have received treatment with no more than three lines of therapy overall in the metastatic setting (including anti-HER2 targeted therapy or chemotherapy) and must have disease progressed on or after, the most recent line of therapy. per RECIST 1.1.

   * Prior radiotherapy, chemotherapy, hormonal therapies are allowed
   * Endocrine therapies will not be considered as previous lines of therapy in the metastatic setting.
   * Prior neo-adjuvant or adjuvant therapy that resulted in relapse within 6 months of the completion of therapy will be considered a line of treatment for metastatic disease.
   * Dose interruptions, delays, pauses during previous therapy, or changes in therapy to manage toxicity will not constitute a new line of therapy provided disease progression did not occur
7. Subject has at least one measurable lesion per RECIST 1.1.
8. Previous adverse events associated with anti-tumor therapy have been recovered to NCI-CTCAE v4.03 Grade ≤1 (except NCI-CTCAE v4.03 Grade ≤2 alopecia, stable sensory neuropathy, or stabilized electrolyte disturbance after fluid transfusion).
9. Subject has life expectancy ≥12 weeks.
10. Subject has no supportive therapy of blood transfusion or growth factor within 4 weeks before randomization and has adequate organ functions as defined below:

    * Absolute Neutrophil count (≥ 1.5 *109/L)
    * Platelets count (≥ 100 *109/L)
    * Hemoglobin (≥ 90 g/L)
    * Serum creatinine (≤1.5 times the upper limit of normal (ULN)) or calculated creatinine clearance (≥50 mL/min) (per Cockcroft-Gault formula; see Appendix 4)
    * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) or direct bilirubin ≤ 1.0 times the upper limit of normal (ULN)AST and ALT ≤2 times the upper limit of normal (ULN), and liver metastasis must be ≤5 times the upper limit of normal (ULN).
    * Cardiac color Doppler LVEF ≥ 50%
11. Subject has a negative test result of pregnancy test at randomization. Women with childbearing potential are promised to take adequate and effective contraceptive measures or abstinence within six months from the start of the study to the end of the study and after the last medication are admitted. Or the women in the study were women with no potential fertility, defined as:

    * Women underwent surgical sterilization (hysterectomy, bilateral ovariectomy or bilateral salpingectomy), or
    * Women ≥ 60 years of age, or
    * Women are in the ages ≥ 40 years old and <60 years old, and have been amenorrhoeic for 12 months with the results of follicle stimulating hormone examination were in the postmenopausal reference range per testing hospital.
12. Subject with good compliance and willing to have the follow-up visits

Exclusion Criteria:

1. Subject has symptomatic, uncontrolled brain or pia mater metastasis. If subject has known and treated brain metastasis, baseline CT or MRI data within 4 weeks prior to randomization are mandatory to be obtained. Subject should have received brain metastasis treatment for at least four weeks before randomization. If subject needs to use steroids for treatment after randomization, the dosage of steroids (<10 mg/day prednisone or equivalent) should be stable before randomization for at least four weeks without relevant neurological symptoms
2. Subject has third interstitial effusion (e.g. massive pleural and ascites) that cannot be controlled by drainage or other means.
3. Subject has local or systemic anti-tumor treatment within 2 weeks prior to randomization, including radiotherapy, chemotherapy, surgical resection (major surgery for breast cancer), or target therapy, and endocrine therapy for anti-tumor within 7 days prior to randomization.
4. Subject has any investigational treatment within 4 weeks prior to randomization (including margetuximab)
5. Subject has history of major surgery with unrecovered surgical effect within 4 weeks prior to randomization.
6. Subject has other malignant tumor (complete cured in situ cervical cancer, cutaneous basal cell carcinoma or cutaneous squamous cell carcinoma are not included) within 5 years prior to randomization.
7. Subject has severe and uncontrolled disease, including but not limited to

   * Uncontrollable nausea and vomiting, and any other severe gastrointestinal disorders
   * Active viral infections, e.g. human immunodeficiency virus (HIV), hepatitis B (HBV; HbsAg positive, HBV-DNA (≥103 copies/ml or (≥500 IU/ml), hepatitis C (HCV) etc.
   * Severe uncontrollable diabetes, hypertension, thyroid diseases etc.
   * Severe uncontrollable pulmonary diseases, e.g. severe contagious pneumonia, interstitial lung disease etc.
   * Myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack within 6 months prior to randomization; clinically significant arrhythmia, congestive heart failure (NYHA II-IV), pericarditis or severe pericardial effusion, myocarditis, etc.
8. Subject has known allergy to recombinant proteins, polysorbide 80, benzyl alcohol or any excipients contained in manufacturing of margetuximab, trastuzumab or other study treatments. For subject with previous transfusion reactions to trastuzumab or other monoclonal antibodies, if there is no contraindication for trastuzumab treatment, the subject is eligible for enrollment.
9. Subject has contraindication of using trastuzumab, or confounding disease that may prevent subject from using chemotherapy prescribe by the investigator.
10. Subject has vaccination with any live virus vaccine within four weeks prior to randomization; inactivated influenza vaccine is allowed.
11. Subject who is pregnant or breastfeeding, or who is expected to be pregnant during the period of the study
12. Dementia or any mental condition may impede understanding and informed consent
13. Any disease, treatment, or laboratory abnormalities that may interfere with the results of the study, affect the subject's full participation in the study, or that the investigator does not consider that the subject is appropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by BICR (RECIST 1.1) | Approximately 18 months after the first subject is randomized; anticipated evaluation Jul 2020.
  the time from randomization date to the date of first documented disease progression or death from any cause, whichever occurs first. The confirmation of disease progression is per RECIST 1.1, and evaluation made by BICR

SECONDARY OUTCOMES:
Overal Survival (OS) | Approximately 15 months after the last subject is randomized
  the time from randomization date to the date of death from any cause
PFS assessed by Investigator | Approximately 18 months
  the time from randomization date to the date of first documented disease progression or death from any cause, whichever occurs first. The confirmation of disease progression is per RECIST 1.1, and evaluation made by investigator
Objective Response Rate (ORR) assessed by BICR | Approximately 18 months
  the proportion of subjects in the response evaluable population achieving a best response of CR or PR when such responses are confirmed 6 weeks after initial observation of response. Subjects who have no assessment will be considered as non-responders
Duration of Response (DoR) assessed by BICR | the time from initial response to date of first documented disease progression or death from any cause, whichever occurs first
  To evaluate the DoR assessed by BICR
Clinical Beneficial Rate (CBR) | Approximately 18 months
  the proportion of subjects in the response evaluable population achieving a best response of CR, PR, or SD
FcγR | at baseline (before first dose of treatment)
  To evaluate the effects of allelic variation in FcγR on the efficacy of margetuximab in all patients receiving study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Zhang Q, Ouyang Q, Li W, Chiu J, Yan M, Lu YS, Sun S, Li H, Du Y, Wang X, Sun T, Yin Y, Wang H, Ye F, Shen K, Wang J, Pan Y, Wang S, Yang J, Wu X, Dai MS, Cheng J, Teng Y, Su F, Wu X, He J, Fu P, Yang L, Xin Y, Wang X, Jiang Z. Efficacy and safety of margetuximab plus chemotherapy vs. trastuzumab plus chemotherapy in Chinese patients with pretreated HER2-positive advanced metastatic breast cancer: results from a randomized, open-label, multicenter, phase II bridging study. Transl Breast Cancer Res. 2022 Oct 31;3:31. doi: 10.21037/tbcr-22-35. eCollection 2022. PMID 38751523